CLINICAL TRIAL: NCT05596903
Title: Effect of Eye Movement Desensitization and Reprocessing Therapy 2.0 Online Group Protocol on Traumatic Experiences Based on Traffic Accident: A Randomized Controlled Trial
Brief Title: Effect of Eye Movement Desensitization and Reprocessing Therapy 2.0 Online Group Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academy of Therapeutic Sciences, Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TBA2021
Record Dates: First submitted 2022-10-21; First posted 2022-10-27 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Post Traumatic Stress Disorder
Keywords: EMDR; Post-traumatic stress disorder; Anxiety; Depression; Stress; Trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Control Group (3) vs EMDR 2.0 Group Intervention (3)
Who Masked: Participant
Masking Description: Single
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMDR 2.0 (Experimental): EMDR 2.0 Online Group protocol will be administered.
  Interventions: Other: EMDR 2.0 group protocol
- Control (Active Comparator): Mental Health Gap Action Programme (mhGAP) will be administered.
  Interventions: Other: Mhgap stress module

INTERVENTIONS:
Other: EMDR 2.0 group protocol — EMDR 2.0 group protocol
  Arms: EMDR 2.0
Other: Mhgap stress module — Mhgap stress module
  Arms: Control

SUMMARY:
In this study, it will be investigated the efficacy of Eye Movement Desensitization and Reprocessing Therapy 2.0 Online Group Protocol on post-traumatic symptoms compared to control group. Therefore, the randomized control trial is based on Eye Movement Desensitization and Reprocessing Therapy 2.0 group as an intervention.

DETAILED DESCRIPTION:
Eye Movement Desensitization and Reprocessing Therapy is an evidence-based psychotherapy approach, and it is proven as efficient in primarily post-traumatic symptom disorder. EMDR 2.0 is a new approach which is used for the cases that are not answering the standard EMDR protocols. According to the recent studies, both EMDR and EMDR 2.0 show a greater decrease in emotionality and vividness in similar time based on session numbers (Matthijssen, 2021). Also, it is found that EMDR 2.0 requires lower set numbers (shorter sessions) compared to EMDR.

In this study, it will be investigated the efficacy of EMDR 2.0 Online Group Protocol on post-traumatic symptoms compared to control group. Therefore, the randomized control trial is based on EMDR 2.0 group as an intervention. Compared to previous EMDR 2.0 individual settings, this study is based on a group protocol made by our team. This group protocol has been tested in a pilot study on volunteer mental health professionals. The results of this pilot study showed that EMDR 2.0 group protocol was successful, and investigators decided to begin the randomized control trial research.

ELIGIBILITY:
Inclusion Criteria:

* Being older than 18
* Having a traffic accident between 6 months and 10 years
* Having necessary knowledge on using relevant technological devices

Exclusion Criteria:

* Having mental deterioration after the accident
* Having a lower score of 7 on Adverse Childhood Experiences (ACEs)
* Having pre-existing psychotic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) | 1-week and 1-month follow-up
  Depression, stress and anxiety scores will significantly change. Scores for depression, anxiety and stress are calculated by summing the scores. The scores are between 0-3, and more scores mean worse results.
  for the relevant items
Impact of Events Scale Revised (IES-R) | 1-week and 1-month follow-up
  Intrusion and hyperarousal scores will significantly change. The maximum mean score on each of the three subscales is '4', therefore the maximum 'total mean' IES- R score is 12. Lower scores are better.

CONTACTS AND LOCATIONS:
Locations (1):
- Academy of Therapeutic Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Baddeley A. Working memory: theories, models, and controversies. Annu Rev Psychol. 2012;63:1-29. doi: 10.1146/annurev-psych-120710-100422. Epub 2011 Sep 27. PMID 21961947
- [Result] de Jongh A, Ernst R, Marques L, Hornsveld H. The impact of eye movements and tones on disturbing memories involving PTSD and other mental disorders. J Behav Ther Exp Psychiatry. 2013 Dec;44(4):477-83. doi: 10.1016/j.jbtep.2013.07.002. Epub 2013 Jul 13. PMID 23892070
- [Result] Littel, M., Remijn, M., Tinga, A. M., Engelhard, I. M., & van den Hout, M. A. (2017). Stress Enhances the Memory-Degrading Effects of Eye Movements on Emotionally Neutral Memories. Clinical Psychological Science, 5(2), 316-324. https://doi.org/10.1177/2167702616687292
- [Result] Littel M, van Schie K. No evidence for the inverted U-Curve: More demanding dual tasks cause stronger aversive memory degradation. J Behav Ther Exp Psychiatry. 2019 Dec;65:101484. doi: 10.1016/j.jbtep.2019.101484. Epub 2019 May 13. PMID 31125845
- [Result] Matthijssen SJMA, Verhoeven LCM, van den Hout MA, Heitland I. Auditory and Visual Memories in PTSD Patients Targeted with Eye Movements and Counting: The Effect of Modality-Specific Loading of Working Memory. Front Psychol. 2017 Nov 3;8:1937. doi: 10.3389/fpsyg.2017.01937. eCollection 2017. PMID 29163311
- [Result] Matthijssen SJMA, van Beerschoten LM, de Jongh A, Klugkist IG, van den Hout MA. Effects of "Visual Schema Displacement Therapy" (VSDT), an abbreviated EMDR protocol and a control condition on emotionality and vividness of aversive memories: Two critical analogue studies. J Behav Ther Exp Psychiatry. 2019 Jun;63:48-56. doi: 10.1016/j.jbtep.2018.11.006. Epub 2018 Nov 27. PMID 30514434
- [Result] Matthijssen SJMA, van Schie K, van den Hout MA. The Effect of modality specific interference on working memory in recalling aversive auditory and visual memories. Cogn Emot. 2019 Sep;33(6):1169-1180. doi: 10.1080/02699931.2018.1547271. Epub 2018 Nov 22. PMID 30465479
- [Result] Matthijssen SJMA, Brouwers T, van Roozendaal C, Vuister T, de Jongh A. The effect of EMDR versus EMDR 2.0 on emotionality and vividness of aversive memories in a non-clinical sample. Eur J Psychotraumatol. 2021 Sep 22;12(1):1956793. doi: 10.1080/20008198.2021.1956793. eCollection 2021. PMID 34567439
- [Result] van den Hout MA, Eidhof MB, Verboom J, Littel M, Engelhard IM. Blurring of emotional and non-emotional memories by taxing working memory during recall. Cogn Emot. 2014;28(4):717-27. doi: 10.1080/02699931.2013.848785. Epub 2013 Nov 7. PMID 24199660
- [Result] van Veen SC, van Schie K, Wijngaards-de Meij LD, Littel M, Engelhard IM, van den Hout MA. Speed Matters: Relationship between Speed of Eye Movements and Modification of Aversive Autobiographical Memories. Front Psychiatry. 2015 Apr 7;6:45. doi: 10.3389/fpsyt.2015.00045. eCollection 2015. PMID 25904871
- [Derived] Yasar AB, Gundogmus I, Kubilay D, Alban Tunca G, Uygun E, Zat Ciftci Z, Kavakci O. The effectiveness of online Eye Movement Desensitization and Reprocessing 2.0 Group Protocol on post-traumatic stress disorders symptoms, depression, anxiety, and stress in individuals who have experienced a traffic accident: a randomized-controlled study. Front Psychiatry. 2025 May 9;16:1452206. doi: 10.3389/fpsyt.2025.1452206. eCollection 2025. PMID 40417270

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT05596903/Prot_SAP_ICF_000.pdf